CLINICAL TRIAL: NCT02405715
Title: Combined Use of Intranasal Oxytocin and Interpersonal Psychotherapy for the Treatment of Major Depressive Disorder (MDD): A Randomized Controlled Trial
Brief Title: Therapy With an Oxytocin Adjunct for Major Depression
Acronym: TOAD2015
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Concordia University, Montreal (Other)
Responsible Party: Principal Investigator, Mark Ellenbogen, Associate Professor, Concordia University, Montreal
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIHR-12678
Record Dates: First submitted 2015-03-02; First posted 2015-04-01 (Estimated); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Spray And Interpersonal Psychotherapy (Placebo Comparator): Participants will receive 6 sprays of a placebo nasal spray prior to the beginning of each session of interpersonal psychotherapy (16 sessions in total).
  Interventions: Drug: Oxytocin nasal spray or placebo
- Oxytocin Spray And Interpersonal Psychotherapy (Experimental): Participants will receive 6 sprays of a oxytocin nasal spray prior to the beginning of each session of interpersonal psychotherapy (16 sessions in total). Each spray will contain 4IU of oxytocin, for a total dose of 24IU.
  Interventions: Drug: Oxytocin nasal spray or placebo

INTERVENTIONS:
Drug: Oxytocin nasal spray or placebo
  Other Names: Syntocinon

SUMMARY:
This study evaluates the addition of intranasal oxytocin to the treatment of Major Depression using interpersonal psychotherapy. Half of the participants will receive a placebo adjunct to interpersonal psychotherapy, and the other half will receive oxytocin.

DETAILED DESCRIPTION:
Depression is a debilitating mental health condition that carries great consequences for both the individual and society. Crucially, at least one third of depressed patients do not respond to existing interventions and relapse rates are high, alerting scientists to the need to explore possible adjunctive treatments and novel therapeutic targets. In this regard, research on the use of oxytocin in the treatment of depression is promising.

It is well documented that interpersonal stress predicts the onset of depression, and that social isolation is a symptom of psychological distress that can leave patients with a poor prognosis for recovery. Therapeutic interventions focused on the alleviation of social conflict and strengthening of social bonds (i.e. Interpersonal Psychotherapy; IPT) show greater efficacy for the treatment of depression than other psychological interventions (NIMH Treatment of Depression Collaborative Research Program; Elkin et al. 1984). It has been posited that oxytocin, a naturally produced hormone that is involved in social-support seeking and stress-regulation, could represent a biological link between social stress and depression in adulthood. The salubrious effect of exogenous oxytocin on human social behavior is well documented: Oxytocin has been shown to make individuals feel more securely attached in their social relationships, increase their trust in others and openness to new ideas, improve their recall of specific and positive social autobiographical memories, and improve social learning. Importantly, these factors have been shown to improve the efficacy of Interpersonal Psychotherapy. Thus, It stands to reason that the use of oxytocin as an adjunct to IPT could improve its efficacy for the treatment of depression, which is an important prospect when considering that a third of patients do not respond to existing therapies.

In the proposed research project, we will conduct a Randomized Controlled Trial for the treatment of Major Depression with IPT and adjunctive oxytocin. Patients will be screened for eligibility, undergo structured psychotherapy for twelve weeks, and will be followed longitudinally for changes in quality of social functioning, interpersonal stress, psychiatric symptoms and depressive relapse. Establishing novel interventions for depression could position healthcare providers to better alleviate the burden and personal suffering caused by this disorder.

ELIGIBILITY:
Inclusion Criteria

• Current Major Depressive Episode

Exclusion Criteria

* Visual impairment
* Major medical illness [A condition that is chronic and associated with impaired functioning, distress, or frequent medical intervention), in particular, subjects with evidence or history of malignancy or any significant hematological, endocrine, cardiovascular (including any rhythm disorder), respiratory, renal, hepatic, or gastrointestinal disease
* Acute or chronic nasal diseases or obstruction
* Current (in the last month) use of any endocrine-relevant or psychotropic medication other than prescription antidepressants
* Current substance dependence or abuse
* Use of illicit drugs (stimulants, narcotics, psychedelics/hallucinogens, non-prescription medication) in the past 8 weeks
* Lifetime history of a psychosis (except if part of MDD) or pervasive developmental disorder
* Past or current comorbid axis-1 disorder except Dysthymia, Adjustment Disorder, Generalized Anxiety Disorder, Social Phobia, and Specific Phobia.
* Female Only: Females of child bearing potential cannot be pregnant or breastfeeding in order to participate in this study. They must not be planning to become pregnant, and must be willing to use appropriate contraception throughout the study.
* Female Only: To control for hormonal changes related to pregnancy, females will also be excluded if they have previously given birth.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Diagnostic status: Major Depressive Episode Using The SCID-IV [Change Score] | Baseline, 4 months later (following therapy)
  Diagnosis of Major Depressive Episode Will Be Diagnosed Using The SCID-IV
Depressive symptoms (clinician-rated) 9Hamilton Rating Scale for Depression (HRS-D)[Change Score] | Baseline, 4 months later (following therapy)
  Hamilton Rating Scale for Depression (HRS-D)
Depressive symptoms (clinician-rated) Inventory for Depressive Symptomology (IDS-C) [Change Score] | Baseline, 4 months later (following therapy)
  Inventory for Depressive Symptomology (IDS-C)
Stress and social functioning (Global Axis of Functioning using the SCID-IV (GAF) [Change Score] | Baseline, 4 months later (following therapy)
  Global Axis of Functioning using the SCID-IV (GAF)
Patient dropout rate [Number of sessions missed] | includes baseline up to 4 months following baseline assessment (until the end of therapy)
  patient dropout rate
Depressive Symptoms (patient-rated) (Beck Depression Inventory-II (BDI-II) [Change Score] | Baseline up to 10 months later (slope of change over time)
Diagnostic status: Major Depressive Episode Using The SCID-IV [Change Score] | 4 months later (following therapy) and 10 months later (6 months following therapy)
  Diagnosis of Major Depressive Episode Will Be Diagnosed Using The SCID-IV
Depressive symptoms (clinician-rated) 9Hamilton Rating Scale for Depression (HRS-D) [Change Score] | 4 months later (following therapy) and 10 months later (6 months following therapy)
  Hamilton Rating Scale for Depression (HRS-D)
Depressive symptoms (clinician-rated) Inventory for Depressive Symptomology (IDS-C) [Change Score] | 4 months later (following therapy) and 10 months later (6 months following therapy)
  Inventory for Depressive Symptomology (IDS-C)
Stress and social functioning (Global Axis of Functioning using the SCID-IV (GAF) [Change Score] | 4 months later (following therapy) and 10 months later (6 months following therapy)
  Global Axis of Functioning using the SCID-IV (GAF)

SECONDARY OUTCOMES:
Stress and social functioning (clinician-rated) (UCLA Life Stress Interview - Chronic Stress Module (UCLA) [Change Score] | Baseline, 4 months later (following therapy)
  UCLA Life Stress Interview - Chronic Stress Module (UCLA)
Biological stress reactivity (Daily Diurnal Cortisol) [Change Score] | Baseline, 4 months later (following therapy)
  Daily Diurnal Cortisol (2 days)
Working alliance (clinician-rated) (Working Alliance Inventory (WAI) [Change Score] | Baseline up to 4 months later (slope of change over time)
  Working Alliance Inventory (WAI)
Social functioning (patient-rated) (Social Adjustment Scale- Self-Report (SAS-SR) + MSPSS) COMPOSITE SCORE [Change Score] | Baseline up to 10 months later (slope of change over time)
  Social Adjustment Scale- Self-Report (SAS-SR) + MSPSS
Stress (patient-rated) (Perceived Stress Scale (PSS) [Change Score] | Baseline up to 10 months later (slope of change over time)
  Perceived Stress Scale (PSS)
Anxiety (patient-rated) (Beck Anxiety Inventory (BAI) [Change Score] | Baseline up to 10 months later (slope of change over time)
  Beck Anxiety Inventory (BAI)
Therapeutic Alliance (patient-rated) (Working Alliance Inventory (WAI) | Baseline up to 4 months later (slope of change over time)
  Working Alliance Inventory (WAI)
Usefulness of Therapy (patient-rated); COMPOSITE SCORE | Baseline up to 4 months later (slope of change over time)
  Measure by score on Helpful Aspects of Therapy (HAT)
Stress and social functioning (clinician-rated) (UCLA Life Stress Interview - Chronic Stress Module (UCLA) [Change Score] | 4 months later (following therapy) and 10 months later (6 months following therapy)
  UCLA Life Stress Interview - Chronic Stress Module (UCLA)
Biological stress reactivity (Daily Diurnal Cortisol) [Change Score] | 4 months later (following therapy) and 10 months later (6 months following therapy)
  Daily Diurnal Cortisol (2 days)

OTHER OUTCOMES:
Moderation by personality (NEO-PI-R) | Baseline
  NEO-PI-R; Moderation by extraversion
Mediation by personality (NEO-PI-R) [Change Score] | Baseline up to 10 months later [Slope of Change]
  NEO-PI-R; Mediation by extraversion
Moderation by attachment (ECR, AAI) [COMPOSITE SCORE] | Baseline
  ECR, AAI: Moderation by attachment style
Moderation by attachment (ECR, AAI) [COMPOSITE SCORE] | Baseline up to 10 months later [Slope of Change]
  ECR, AAI: Mediation by attachment style
Adverse Events [Average Score] COMPOSITE | baseline up to 4 months
  In-house measure of adverse events weekly

CONTACTS AND LOCATIONS:
Locations (1):
- Concordia University, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Ellenbogen MA, Cardoso C, Serravalle L, Vadaga K, Joober R. The effects of intranasal oxytocin on the efficacy of psychotherapy for major depressive disorder: a pilot randomized controlled trial. Psychol Med. 2024 Jul;54(9):2122-2132. doi: 10.1017/S0033291724000217. Epub 2024 Mar 6. PMID 38445382